CLINICAL TRIAL: NCT01736969
Title: Microcyn Scar Management HydroGel, K103163 vs. Kelo-cote® Scar Gel for the Management of Hypertrophic or Keloid Scars
Brief Title: A Substantial Equivalence Study of RD04723 and Predicate Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oculus Innovative Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSM-RD-023
Record Dates: First submitted 2012-10-12; First posted 2012-11-29 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Hypertrophic Scar; Keloid Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic; Keloid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- RD047-023 (Experimental): RD-047-023
  Interventions: Device: RD047-023
- Predicate Device (Active Comparator): legally marketed predicate device
  Interventions: Device: Predicate Device

INTERVENTIONS:
Device: RD047-023 — Experimental hydrogel
  Arms: RD047-023
Device: Predicate Device
  Other Names: Kelo-Cote
  Arms: Predicate Device

SUMMARY:
The purpose of this study is to determine whether a developmental formulation is substantially equivalent to the predicate device in the treatment of hypertrophic and keloid scars.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent and release health information
* Ability to follow study instructions and study requirements
* Have a hypertrophic or keloid scar accessible for treatment and evaluation
* Negative pregnancy test for women of childbearing potential
* Agreement to use effective birth control method for study duration

Exclusion Criteria:

* History of allergy or sensitivity to components
* History of diabetes
* History of collagen vascular disorders
* Anticipated need for surgery or hospitalization during the study
* Pregnant, nursing, or planning a pregnancy during the study
* Current enrollment in an investigational drug or device study or participation in such a study within the last 30 days prior to Baseline (Day 0)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Comparison between groups in Vancouver Scar Scale total score from Baseline to Day 112 (or early termination) | 4 weeks, 8 weeks, 12 weeks
  Vascularity, height/thickness, pliability, and pigmentation. Scoring from zero to thirteen.

SECONDARY OUTCOMES:
Pain and itch | 4 weeks, 8 weeks, 12 weeks
  Patient assessment of pain and itch. Scoring from 0-3.
Adverse Events | Baseline, Weeks: 2, 4, 8, 12 and early termination
  Number of subjects with related adverse events
Treatment satisfaction | 8 weeks, 12 weeks
  Patient assessment (satisfaction) with scar treatment. Stated as: "very good, good, moderate or unsatisfactory".

CONTACTS AND LOCATIONS:
Overall Officials: Janet C DuBois, MD, Principal Investigator — Derm Research, PLLC
Locations (1):
- DermResearch Inc, Austin, Texas, United States